CLINICAL TRIAL: NCT04989790
Title: Clinical Effectiveness of the "PICU Up!" Multifaceted Early Mobility Intervention for Critically Ill Children: A Pragmatic, Stepped-wedge Trial
Brief Title: Clinical Effectiveness of the "PICU Up!" Multifaceted Early Mobility Intervention for Critically Ill Children
Acronym: PICU Up!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00297110; R01HD103811 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Child; Intensive Care Unit Acquired Weakness; Critical Illness; Hospital Acquired Pressure Ulcer
Keywords: physical rehabilitation; post-intensive care syndrome; pediatric intensive care unit; sleep; sedation; delirium; physical therapy; occupational therapy
MeSH Terms: conditions — Critical Illness; postintensive care syndrome; Delirium

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline/Pre-implementation (No Intervention): Usual PICU care
- Intervention/Post-implementation (Active Comparator): PICU Up! is a multifaceted, inter-professional pathway that is integrated into routine PICU practice to safely optimize early and progressive patient mobility.
  Interventions: Other: PICU Up!

INTERVENTIONS:
Other: PICU Up! — PICU Up! incorporates the screening process for determining a patient's appropriate activity level into the daily rounding workflow for all PICU patients, with a tiered activity plan based on clinical parameters to individualize goals based on each child's unique needs. While the patient's PICU Up! level is based on objective criteria, the interprofessional team collectively determines the daily activity goal(s) through shared decision-making which is documented in the medical record on morning rounds. The intervention facilitates daily discussion of 1) analgesia; 2) extubation readiness testing; 3) sedation level and goal; 4) delirium screening and management; 5) mobility goal including physical and occupational therapy consultation by PICU Day 3; 6) sleep promotion; and 7) family engagement in mobility.
  Arms: Intervention/Post-implementation

SUMMARY:
While mortality in U.S. pediatric intensive care units (PICUs) is improving, surviving children frequently develop persistent physical, cognitive, and psychological impairments. Over half of critically ill children experience potentially preventable PICU-acquired morbidities, with mechanically ventilated children being at greatest risk. In critically ill adults, randomized trials have shown that progressive mobility, started early (within 3 days of initiating mechanical ventilation), decreases muscle weakness and the duration of mechanical ventilation. However, similar randomized studies have not been conducted in the PICU. The investigator's prior studies revealed that less than 10 percent of critically ill children at the highest risk of functional decline are evaluated by a physical or occupational therapist within 3 days of PICU admission. Given the interplay of sedation, delirium, sleep, and immobility in the PICU, single-component interventions, such as sedation protocolization, have not consistently shown benefit for decreasing mechanical ventilation duration. Thus, the investigators developed the first pediatric-specific, interprofessional intervention (PICU Up!) to integrate goal-directed sedation, delirium prevention, sleep promotion, and family engagement into daily PICU care in order to facilitate early and progressive mobility. The investigators have demonstrated the safety and feasibility of this pragmatic, multifaceted strategy in both single-site and multicenter pilot studies. Hence, the next phase of the investigators research is to evaluate the clinical effectiveness and delivery of the PICU Up! intervention across a range of PICU patients and health systems. The investigators propose a pragmatic, stepped-wedge, cluster randomized controlled trial that will include 10 academic and community hospitals in the United States, with the following Aims: 1) Evaluate if the PICU Up! intervention, delivered under real-world conditions, decreases mechanical ventilation duration (primary outcome) and improves delirium and functional status compared to usual care in critically ill children; and 2) Conduct a multi-stakeholder, mixed-methods process evaluation to identify key contextual factors associated with delivery of PICU Up!. If proven effective, the PICU Up! intervention has potential to profoundly change medical care in the PICU and substantially impact public health by improving outcomes for the growing number of pediatric survivors of critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation via oral or nasal endotracheal tube ≥ 48 hours at 7 a.m. on PICU Day 3

Exclusion Criteria:

* Active or anticipated withdrawal of life support within 48 hours
* Open chest or open abdomen
* Current use of Extracorporeal Membrane Oxygenation (ECMO)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1440 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation | Through Day 21
  In computing duration of mechanical ventilation, the investigators will consider Time 0 as the time of endotracheal intubation or PICU admission for patients intubated at an outside hospital, and continuing until the first time the endotracheal tube was continuously absent for at least 24 hours. Patients will be assigned 21 days for ventilation duration if they remain intubated and mechanically ventilated, are transferred to another facility while ventilated or die prior to day 21 without ever remaining off mechanical ventilation ventilation (via endotracheal tube) for more than 24 continuous hours. If a patient is transitioned to mechanical ventilation via a new tracheostomy those days will be counted as mechanical ventilation days.

SECONDARY OUTCOMES:
Proportion of Days with Delirium | Through Day 21
  Defined as the number of days with delirium divided by the total number of days that the child is at risk for delirium (i.e. the number of days that the patient is in the PICU and free of coma and therefore assessable for delirium).
Change in Functional Status as assessed by the Pediatric Cerebral Performance Category (PCPC) scale | Through Day 21
  The Pediatric Cerebral Performance Category is a global scale based on observer impressions. It's is a six point graded scale of increasing disability from 1 normal function, to 6 death. Scores include 1 for good, 2 for mild disability, 3 for moderate disability, 4 for severe disability, and 5 for vegetative state or coma. Higher scores indicating worse performance or functional morbidity.
Change in Functional Status as assessed by the Pediatric Overall Performance Category (POPC) scale | Through Day 21
  The Pediatric Overall Performance Category (POPC) is a global scale based on observer impressions. It's is a six point graded scale of increasing disability from 1 normal function, to 6 death. Scores include 1 for good, 2 for mild disability, 3 for moderate disability, 4 for severe disability, and 5 for vegetative state or coma. Higher scores indicating worse performance or functional morbidity.

OTHER OUTCOMES:
PICU length of stay | Through Day 21
  PICU length of stay days
Percentage of patients PICU mortality | Through Day 21
  PICU mortality
Number of patients discharged to home | Through Day 21
  Number of patients discharged to home
Number of patients discharged to inpatient floor | Through Day 21
  Number of patients discharged to inpatient floor
Number of patients discharged to inpatient rehabilitation | Through Day 21
  Number of patients discharged to inpatient rehabilitation
Number of patients discharged to other hospital | Through Day 21
  Number of patients discharged to other hospital
Percentage of patients with new pressure injuries | Through Day 21
  Percentage of patients with new pressure injuries
Percentage of patients with physical therapy consultation | Day 3
  Physical therapy consultation by PICU
Percentage of patients with occupational therapy consultation | Day 3
  Occupational therapy consultation by PICU
Mean daily Opioid exposure | Through Day 21
  Opioid exposure: mean daily morphine and equivalents (mg/kg/day) via chart review
Mean daily Benzodiazepine exposure | Through Day 21
  Benzodiazepine exposure: mean daily benzodiazepine equivalents (mg/kg/day) via chart review

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Kudchadkar, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - Valley Children's Hospital, Madera, California
  - Nemours Children's Hospital of the Nemours Foundation, Orlando, Florida
  - Norton Children's Hospital: University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Hennepin Healthcare: University of Minnesota, Minneapolis, Minnesota
  - Children's Hospital at Dartmouth: Geisel School of Medicine, Lebanon, New Hampshire
  - UNC Children's: University of North Carolina, Chapel Hill, North Carolina
  - Janet Weis Children's Hospital: Geisinger Commonwealth School of Medicine, Danville, Pennsylvania
  - Texas Children's Hospital: Baylor College of Medicine, Houston, Texas
  - West Virginia University Medicine Children's: West Virginia University, Morgantown, West Virginia
  - Children's Hospital of Wisconsin: Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
Data generated in this grant will be presented in a timely fashion at national and international meetings and in publications. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive PubMed Central. The investigators plan to share data from this research with other researchers who have interests in improving outcomes in critically ill children through early and progressive mobility interventions. Written proposals for data sharing requests will be accepted and reviewed by an independent review committee to ensure the proposal is scientifically and methodologically sound and not duplicative with other analyses. If approved, data sharing would occur after establishing a data use agreement with institutional signing authorities of each institution. Medical record and outcomes data will then be made available in the form of deidentified datasets with no identifiers in keeping with NIH Data Sharing Policy and Implementation Guidance.

REFERENCES:
- [Background] Wieczorek B, Ascenzi J, Kim Y, Lenker H, Potter C, Shata NJ, Mitchell L, Haut C, Berkowitz I, Pidcock F, Hoch J, Malamed C, Kravitz T, Kudchadkar SR. PICU Up!: Impact of a Quality Improvement Intervention to Promote Early Mobilization in Critically Ill Children. Pediatr Crit Care Med. 2016 Dec;17(12):e559-e566. doi: 10.1097/PCC.0000000000000983. PMID 27759596
- [Background] Patel RV, Redivo J, Nelliot A, Eakin MN, Wieczorek B, Quinn J, Gurses AP, Balas MC, Needham DM, Kudchadkar SR. Early Mobilization in a PICU: A Qualitative Sustainability Analysis of PICU Up! Pediatr Crit Care Med. 2021 Apr 1;22(4):e233-e242. doi: 10.1097/PCC.0000000000002619. PMID 33315754
- [Background] Kudchadkar SR, Nelliot A, Awojoodu R, Vaidya D, Traube C, Walker T, Needham DM; Prevalence of Acute Rehabilitation for Kids in the PICU (PARK-PICU) Investigators and the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Physical Rehabilitation in Critically Ill Children: A Multicenter Point Prevalence Study in the United States. Crit Care Med. 2020 May;48(5):634-644. doi: 10.1097/CCM.0000000000004291. PMID 32168030
- [Background] Choong K, Canci F, Clark H, Hopkins RO, Kudchadkar SR, Lati J, Morrow B, Neu C, Wieczorek B, Zebuhr C. Practice Recommendations for Early Mobilization in Critically Ill Children. J Pediatr Intensive Care. 2018 Mar;7(1):14-26. doi: 10.1055/s-0037-1601424. Epub 2017 Apr 10. PMID 31073462
- [Background] Traube C, Silver G, Reeder RW, Doyle H, Hegel E, Wolfe HA, Schneller C, Chung MG, Dervan LA, DiGennaro JL, Buttram SD, Kudchadkar SR, Madden K, Hartman ME, deAlmeida ML, Walson K, Ista E, Baarslag MA, Salonia R, Beca J, Long D, Kawai Y, Cheifetz IM, Gelvez J, Truemper EJ, Smith RL, Peters ME, O'Meara AM, Murphy S, Bokhary A, Greenwald BM, Bell MJ. Delirium in Critically Ill Children: An International Point Prevalence Study. Crit Care Med. 2017 Apr;45(4):584-590. doi: 10.1097/CCM.0000000000002250. PMID 28079605
- [Background] Walker TC, Kudchadkar SR. Early mobilization in the pediatric intensive care unit. Transl Pediatr. 2018 Oct;7(4):308-313. doi: 10.21037/tp.2018.09.02. PMID 30460183
- [Background] Hopkins RO, Choong K, Zebuhr CA, Kudchadkar SR. Transforming PICU Culture to Facilitate Early Rehabilitation. J Pediatr Intensive Care. 2015 Dec;4(4):204-211. doi: 10.1055/s-0035-1563547. PMID 27134761
- [Background] Ista E, Scholefield BR, Manning JC, Harth I, Gawronski O, Bartkowska-Sniatkowska A, Ramelet AS, Kudchadkar SR; EU PARK-PICU Collaborators. Mobilization practices in critically ill children: a European point prevalence study (EU PARK-PICU). Crit Care. 2020 Jun 24;24(1):368. doi: 10.1186/s13054-020-02988-2. PMID 32576273
- [Background] Wieczorek B, Burke C, Al-Harbi A, Kudchadkar SR. Early mobilization in the pediatric intensive care unit: a systematic review. J Pediatr Intensive Care. 2015;2015(4):129-170. doi: 10.1055/s-0035-1563386. Epub 2015 Sep 3. PMID 26380147
- [Background] Flaigle MC, Ascenzi J, Kudchadkar SR. Identifying Barriers to Delirium Screening and Prevention in the Pediatric ICU: Evaluation of PICU Staff Knowledge. J Pediatr Nurs. 2016 Jan-Feb;31(1):81-4. doi: 10.1016/j.pedn.2015.07.009. Epub 2015 Sep 9. PMID 26362671
- [Background] Kudchadkar SR, Aljohani O, Johns J, Leroux A, Alsafi E, Jastaniah E, Gottschalk A, Shata NJ, Al-Harbi A, Gergen D, Nadkarni A, Crainiceanu C. Day-Night Activity in Hospitalized Children after Major Surgery: An Analysis of 2271 Hospital Days. J Pediatr. 2019 Jun;209:190-197.e1. doi: 10.1016/j.jpeds.2019.01.054. Epub 2019 Mar 15. PMID 30885646
- [Background] Miura S, Wieczorek B, Lenker H, Kudchadkar SR. Normal Baseline Function Is Associated With Delayed Rehabilitation in Critically Ill Children. J Intensive Care Med. 2020 Apr;35(4):405-410. doi: 10.1177/0885066618754507. Epub 2018 Jan 22. PMID 29357778
- [Background] Choong K, Zorko DJ, Awojoodu R, Ducharme-Crevier L, Fontela PS, Lee LA, Guerguerian AM, Garcia Guerra G, Krmpotic K, McKelvie B, Menon K, Murthy S, Sehgal A, Weiss MJ, Kudchadkar SR. Prevalence of Acute Rehabilitation for Kids in the PICU: A Canadian Multicenter Point Prevalence Study. Pediatr Crit Care Med. 2021 Feb 1;22(2):181-193. doi: 10.1097/PCC.0000000000002601. PMID 33116069
- [Background] Kudchadkar SR, Yaster M, Punjabi NM. Sedation, sleep promotion, and delirium screening practices in the care of mechanically ventilated children: a wake-up call for the pediatric critical care community*. Crit Care Med. 2014 Jul;42(7):1592-600. doi: 10.1097/CCM.0000000000000326. PMID 24717461
- [Background] Ghafoor S, Fan K, Williams S, Brown A, Bowman S, Pettit KL, Gorantla S, Quillivan R, Schwartzberg S, Curry A, Parkhurst L, James M, Smith J, Canavera K, Elliott A, Frett M, Trone D, Butrum-Sullivan J, Barger C, Lorino M, Mazur J, Dodson M, Melancon M, Hall LA, Rains J, Avent Y, Burlison J, Wang F, Pan H, Lenk MA, Morrison RR, Kudchadkar SR. Beginning Restorative Activities Very Early: Implementation of an Early Mobility Initiative in a Pediatric Onco-Critical Care Unit. Front Oncol. 2021 Mar 8;11:645716. doi: 10.3389/fonc.2021.645716. eCollection 2021. PMID 33763377
- [Background] Denlinger K, Young DL, Beier M, Friedman M, Quinn J, Hoyer EH, Kudchadkar SR. Psychometric Testing of the Activity Measure for Post-Acute Care (AM-PAC) in the Pediatric Acute Care Setting. Pediatr Phys Ther. 2021 Jul 1;33(3):149-154. doi: 10.1097/PEP.0000000000000807. PMID 34086622
- [Background] Fayed N, Cameron S, Fraser D, Cameron JI, Al-Harbi S, Simpson R, Wakim M, Chiu L, Choong K. Priority Outcomes in Critically Ill Children: A Patient and Parent Perspective. Am J Crit Care. 2020 Sep 1;29(5):e94-e103. doi: 10.4037/ajcc2020188. PMID 32869071
- [Background] Treble-Barna A, Beers SR, Houtrow AJ, Ortiz-Aguayo R, Valenta C, Stanger M, Chrisman M, Orringer M, Smith CM, Pollon D, Duffett M, Choong K, Watson RS, Kochanek PM, Fink EL; PICU-Rehabilitation Study Group, Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network, and Prevalence of Acute critical Neurological disease in children: A Global Epidemiological Assessment (PANGEA) Investigators. PICU-Based Rehabilitation and Outcomes Assessment: A Survey of Pediatric Critical Care Physicians. Pediatr Crit Care Med. 2019 Jun;20(6):e274-e282. doi: 10.1097/PCC.0000000000001940. PMID 30946294
- [Background] Merritt C, Menon K, Agus MSD, Choong K, McNally D, O'Hearn K, Watson RS, Wong HR, Duffett M, Wypij D, Zimmerman JJ. Beyond Survival: Pediatric Critical Care Interventional Trial Outcome Measure Preferences of Families and Healthcare Professionals. Pediatr Crit Care Med. 2018 Feb;19(2):e105-e111. doi: 10.1097/PCC.0000000000001409. PMID 29394234
- [Background] Choong K, Fraser D, Al-Harbi S, Borham A, Cameron J, Cameron S, Cheng J, Clark H, Doherty T, Fayed N, Gorter JW, Herridge M, Khetani M, Menon K, Seabrook J, Simpson R, Thabane L. Functional Recovery in Critically Ill Children, the "WeeCover" Multicenter Study. Pediatr Crit Care Med. 2018 Feb;19(2):145-154. doi: 10.1097/PCC.0000000000001421. PMID 29394221
- [Background] Ames SG, Alessi LJ, Chrisman M, Stanger M, Corboy D, Sinha A, Fink EL. Development and Implementation of Pediatric ICU-based Mobility Guidelines: A Quality Improvement Initiative. Pediatr Qual Saf. 2021 May 19;6(3):e414. doi: 10.1097/pq9.0000000000000414. eCollection 2021 May-Jun. PMID 34046543
- [Background] Betters KA, Hebbar KB, Farthing D, Griego B, Easley T, Turman H, Perrino L, Sparacino S, deAlmeida ML. Development and implementation of an early mobility program for mechanically ventilated pediatric patients. J Crit Care. 2017 Oct;41:303-308. doi: 10.1016/j.jcrc.2017.08.004. Epub 2017 Aug 9. PMID 28821360
- [Derived] Azamfirei R, Mennie C, Dinglas VD, Fatima A, Colantuoni E, Gurses AP, Balas MC, Needham DM, Kudchadkar SR; on behalf of the PICU Up! Investigators. Impact of a multifaceted early mobility intervention for critically ill children - the PICU Up! trial: study protocol for a multicenter stepped-wedge cluster randomized controlled trial. Trials. 2023 Mar 15;24(1):191. doi: 10.1186/s13063-023-07206-2. PMID 36918956
- See also: NIH Reporter Record of PICU Up! Trial — https://reporter.nih.gov/search/-TyQWv1coE2q0PsxZLOP-Q/project-details/10097465